CLINICAL TRIAL: NCT06889623
Title: Impact of Immediate Cisplatin/Gemcitabine Chemotherapy Following Resection for High-Risk Non-Muscle-Invasive Bladder Cancer: an Open-label, Single-arm, Prospective Trial
Brief Title: Immediate Chemotherapy Following Resection for High-Risk Non-Muscle-Invasive Bladder Cancer
Acronym: HIGCrecur
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Shuxiong Zeng, A.P, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-Urology-NAC-001
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: NMIBC
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immediate GC chemotherapy infusion (Experimental): For enrolled patients receiving immediate cisplatin/gemcitabine chemotherapy via intravenous infusion within 24 hours post transurethral resection of bladder tumor (TURBT), fluid samples were collected before and after TURBT, as well as post-chemotherapy, for UroCAD testing to assess chromosomal instability status and evaluate postoperative tumor residual changes. Subsequently, following EAU guidelines, patients were administered 1 year of intravesical Bacillus Calmette-Guérin (BCG) induction and maintenance therapy, with regular imaging studies and cystoscopic examinations for follow-up to assess the patients' pathological response status.
  Interventions: Procedure: Immediate postoperative chemotherapy

INTERVENTIONS:
Procedure: Immediate postoperative chemotherapy — Systemic chemotherapy with cisplatin/gemcitabine intravenous infusion within 24 hours after TURBT

SUMMARY:
Residual tumors after transurethral resection of bladder tumors (TURBT) range from 17-70%, and floating tumor cells from traditional segmental resection may lead to recurrence if they re-implant in the bladder wall. Immediate systemic chemotherapy post-surgery aims to eliminate microlesions promptly and minimize recurrence risk, yet its safety and efficacy require further exploration. This prospective, single-arm study delves into evaluating the efficacy and safety of immediate postoperative systemic chemotherapy in patients with suspected high-risk non-muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
Bladder cancer ranks as the ninth most prevalent cancer globally, with urothelial carcinoma being the primary form, leading to over 220,000 deaths annually. While 70-75% of bladder cancer cases initially present as non-muscle invasive bladder cancer (NMIBC) with favorable prognoses, the recurrence rate can reach 78% within five years post-standard treatment. The primary objective of transurethral resection of bladder tumors (TURBT) is to accurately diagnose and completely eliminate all visible lesions, as the quality of resection significantly impacts prognosis. However, a systematic review reveals a notable risk of residual tumor post-initial resection. For individuals with high-risk non-muscle invasive bladder cancer (NMIBC), EAU guidelines recommend a follow-up resection 2-6 weeks later. Clinical trials have demonstrated that administering a single chemotherapy session within 24 hours of the initial resection can lower recurrence rates. This approach may work by eradicating floating tumor cells, ablating residual tumor cells, and addressing overlooked small tumors. Gemcitabine and cisplatin (GC) have good efficacy and tolerance in patients with bladder cancer and have become the most commonly used regimen in the neoadjuvant treatment of bladder cancer. There is currently a lack of strong evidence that GC chemotherapy 24 hours after surgery can safely and effectively reduce the risk of recurrence in suspected high-risk NMIBC cases. Our goal is to conduct a prospective clinical trial to investigate the feasibility of this treatment method by evaluating the incidence of adverse events and recurrence-free survival in this group of patients by administering systemic chemotherapy 24 hours after TURBT for patients with suspected high-recurrence bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history and cystoscopy results indicating high-risk NMIBC:

  * High-grade T1
  * Any recurrent high-grade Ta
  * High-grade Ta & Tumor diameter greater than 3 cm or multifocal
  * Any CIS
  * Any BCG failure in patients with high-grade disease
  * Any variant histology
  * Any LVI
  * Any high-grade prostatic urethral involvement
* Patients in generally good condition with a follow-up period of 2 years

Exclusion Criteria:

* Bladder cancer other than UC
* MIBC or benign diseases
* Incomplete tumor resection
* Active infection
* Concurrent upper urinary tract or prostatic urethral UC
* Previous systemic chemotherapy, immunotherapy, or radiotherapy
* Leukopenia/thrombocytopenia
* Serum creatinine greater than twice the normal level
* Uncontrollable urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
One-year recurrence-free survival rate | About two years after the first immediate chemotherapy
  The percentage of patients who remain cancer-free for one year after treatment.

SECONDARY OUTCOMES:
Pathological downstaging rate | About 2-6 weeks after the first immediate chemotherapy
  The percentage of patients whose cancer has decreased in stage following treatment.
The incidence of grade ≥ 3 adverse events（AEs） | About two years after the first immediate chemotherapy
  The frequency of severe or serious side effects experienced by patients during a clinical trial or medical treatment(CTCAE V5.0 ).
UroCAD.MRD Index | TURBT perioperative period, about 15 days
  Body fluid samples were collected from patients before and after TUBRT and chemotherapy for chromosomal instability testing, and the residual tumor status of patients was analyzed by analyzing the changes in the UroCAD.MRD index.

CONTACTS AND LOCATIONS:
Overall Officials: Shuxiong Zeng, M.D. Ph.D, Principal Investigator — Department of Urology, Changhai Hospital, Naval Medical University, Shanghai, China
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babjuk M, Burger M, Capoun O, Cohen D, Comperat EM, Dominguez Escrig JL, Gontero P, Liedberg F, Masson-Lecomte A, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Seisen T, Soukup V, Sylvester RJ. European Association of Urology Guidelines on Non-muscle-invasive Bladder Cancer (Ta, T1, and Carcinoma in Situ). Eur Urol. 2022 Jan;81(1):75-94. doi: 10.1016/j.eururo.2021.08.010. Epub 2021 Sep 10. PMID 34511303
- [Background] Flaig TW, Tangen CM, Daneshmand S, Alva AS, Lucia MS, McConkey DJ, Theodorescu D, Goldkorn A, Milowsky MI, Bangs R, MacVicar GR, Bastos BR, Fowles JS, Gustafson DL, Plets M, Thompson IM Jr, Lerner SP. Long-term Outcomes from a Phase 2 Study of Neoadjuvant Chemotherapy for Muscle-invasive Bladder Cancer (SWOG S1314; NCT02177695). Eur Urol. 2023 Sep;84(3):341-347. doi: 10.1016/j.eururo.2023.06.014. Epub 2023 Jul 4. PMID 37414705
- [Background] Bosschieter J, Nieuwenhuijzen JA, van Ginkel T, Vis AN, Witte B, Newling D, Beckers GMA, van Moorselaar RJA. Value of an Immediate Intravesical Instillation of Mitomycin C in Patients with Non-muscle-invasive Bladder Cancer: A Prospective Multicentre Randomised Study in 2243 patients. Eur Urol. 2018 Feb;73(2):226-232. doi: 10.1016/j.eururo.2017.06.038. Epub 2017 Jul 10. PMID 28705539
- [Background] Pfister C, Gravis G, Flechon A, Chevreau C, Mahammedi H, Laguerre B, Guillot A, Joly F, Soulie M, Allory Y, Harter V, Culine S; VESPER Trial Investigators. Perioperative dose-dense methotrexate, vinblastine, doxorubicin, and cisplatin in muscle-invasive bladder cancer (VESPER): survival endpoints at 5 years in an open-label, randomised, phase 3 study. Lancet Oncol. 2024 Feb;25(2):255-264. doi: 10.1016/S1470-2045(23)00587-9. Epub 2023 Dec 21. PMID 38142702
- [Background] Messing EM, Tangen CM, Lerner SP, Sahasrabudhe DM, Koppie TM, Wood DP Jr, Mack PC, Svatek RS, Evans CP, Hafez KS, Culkin DJ, Brand TC, Karsh LI, Holzbeierlein JM, Wilson SS, Wu G, Plets M, Vogelzang NJ, Thompson IM Jr. Effect of Intravesical Instillation of Gemcitabine vs Saline Immediately Following Resection of Suspected Low-Grade Non-Muscle-Invasive Bladder Cancer on Tumor Recurrence: SWOG S0337 Randomized Clinical Trial. JAMA. 2018 May 8;319(18):1880-1888. doi: 10.1001/jama.2018.4657. PMID 29801011